CLINICAL TRIAL: NCT03316911
Title: MKit: A Pilot Study Testing a Life Skills Application to Address Interpersonal Relationships in College
Brief Title: A Pilot Study Testing a Life Skills Application to Address Interpersonal Relationships in College
Acronym: MKit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Michigan Department of State Police (Unknown)
Responsible Party: Principal Investigator, Michelle Munro-Kramer, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00133004; KL2TR000434 (NIH); KL2TR002241 (NIH); CSA-16-17 (Other: Michigan Department of State Police, Grants and Community Services Division)
Record Dates: First submitted 2017-10-17; First posted 2017-10-23 (Actual); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Sexual Violence; Primary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MKit WebApp Intervention (Experimental): The intervention arm will receive the usual standard of care training package for incoming students at the University of Michigan which includes: 1) Haven, an online module about healthy relationships and sexual violence completed before coming to campus; 2) Relationship Remix, an interactive peer-delivered program on healthy relationships and sexual violence; and 3) Change it Up, a bystander intervention educational theater performance delivered by student actors. In addition, they will receive access the MKit WebApp, which will give them access to content, goal setting, and resources for 14 topic areas.
  Interventions: Behavioral: MKit
- Standard of Care (No Intervention): The control arm will receive the usual standard of care training package for incoming students at the University of Michigan which includes: 1) Haven, an online module about healthy relationships and sexual violence completed before coming to campus; 2) Relationship Remix, an interactive peer-delivered program on healthy relationships and sexual violence; and 3) Change it Up, a bystander intervention educational theater performance delivered by student actors.

INTERVENTIONS:
Behavioral: MKit — MKit is a web-based application that uses a life-skills approach to address healthy relationships and sexual violence. It includes 14 tiles which incorporate information, goal setting, and resources.
  Arms: MKit WebApp Intervention

SUMMARY:
This study utilizes implementation science principles to culturally adapt a pre-existing web-based application (WebApp) for use with college students. The ADAPT-ITT process will be utilized to adapt the WebApp to a diverse (race, ethnicity, gender/sexual identity) college population with a focus on life skills and holistic self-care as reinforcement to currently available primary prevention programming available to incoming students. The study hypothesis is that the adapted WebApp will be usable, acceptable, and students will be willing to use it as a reinforcement to current university primary prevention programming. The study team will also monitor retention of participants over the academic year.

ELIGIBILITY:
Inclusion Criteria:

1. Currently enrolled as a student at the participating university (University of Michigan)
2. Age 18 or older
3. Willing to participate in the study
4. Able to speak and read English
5. Participated in Relationship Remix at Alice Lloyd Hall or Mosher-Jordan Hall during the Fall of 2017. These residence halls were selected due to their similar sizes and demographic populations to allow for "approximate matching" between the control and intervention group.

Exclusion Criteria:

1. Did not complete the Relationship Remix session

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2017-10-22 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Munro-Kramer, PhD,CNM,FNP, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the mandatory primary prevention training sessions, Relationship Remix, offered to all incoming students at the University of Michigan. We specifically recruited in October 22, 2017 - November 17, 2017 from Alice Lloyd Residence Hall (control) and Mosher Jordan Residence Hall (intervention).
Period: Overall Study
Arm/Group | MKit WebApp Intervention | Standard of Care
Started | 122 (2 did not complete baseline survey) | 139 (3 did not complete baseline survey)
3-Month Follow-up Survey | 93 | 112
5-Month Follow-up Survey | 89 | 110
Completed | 89 | 110
Not Completed | 33 | 29
Not completed — Lost to Follow-up | 33 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MKit WebApp Intervention | Standard of Care | Total
Number analyzed (Participants) | 122 | 139 | 261
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.13 (.545) | 18.20 (.554) | 18.17 (.550)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 40 | 56 | 96
  Female | 81 | 80 | 161
  Genderqueer/Gender Nonconforming | 1 | 2 | 3
  Trans Female/Trans Woman | 0 | 1 | 1
  Trans Male/Trans Man | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 72 | 95 | 167
  Black or African American | 3 | 4 | 7
  Hispanic/Latino/Spanish | 6 | 6 | 12
  American Indian/Alaska Native | 1 | 0 | 1
  Asian | 31 | 26 | 57
  Multiple Ethnicity/Other | 9 | 3 | 12
  Middle East/North African | 0 | 4 | 4
  Native Hawaiian/Other Pacific Islander | 0 | 1 | 1
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual or Straight | 102 | 119 | 221
  Gay or Lesbian | 1 | 7 | 8
  Bisexual | 8 | 8 | 16
  Something Else | 4 | 3 | 7
  Prefer not to disclose | 7 | 2 | 9
Year in School [Count of Participants; unit: Participants]
  Freshman | 115 | 132 | 247
  Sophomore | 6 | 5 | 11
  Junior | 0 | 1 | 1
  Senior | 0 | 1 | 1
  Graduate or Professional Student | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: 3-Month Usability
Description: The 10-item System Usability Scale will be used to evaluate the usability of WebApp in the intervention group only. The System Usability Scale (Brook, 1996) includes 10 items that are rated from 1 (Strongly Disagree) to 5 (Strongly Agree). To get a final score the: 1) First, one is subtracted from the score of the odd items; 2) Second, the responses are subtracted from 5 for the even-numbered items; 3) Then the responses are summed and multiplied by 2.5 to get a range of 0-100. A score above 68 is considered above average.
Time Frame: 3-months
Population: Only intervention participants were asked the items on the System Usability Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention
Number analyzed (Participants) | 93
score on a scale | 67.66 (14.87)

2. Primary Outcome: 5-Month Usability
Description: as for outcome 1
Time Frame: 5-months
Population: Only intervention participants were asked the items on the System Usability Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention
Number analyzed (Participants) | 89
score on a scale | 68.88 (14.86)

3. Primary Outcome: 3-Month Acceptability
Description: The 5-item System Acceptability Scale (investigator created) will be used to evaluate the acceptability of the WebApp in the intervention group only. An investigator-created acceptability scale with 5-items will be used to measure acceptability. Four items are scored from 1 (Strongly Agree/Very Likely) to 5 (Strongly Disagree/Very Unlikely) and will be reverse coded. One item assess the frequency of use of the WebApp from 1 (Never) to 5 (Multiple times a week). All five items will be summed for a total score. Scores range from 5-25, with higher scores indicating greater acceptability.
Time Frame: 3-months
Population: Only intervention participants were asked the items on the System Acceptability Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention
Number analyzed (Participants) | 93
score on a scale | 15.53 (3.14)

4. Primary Outcome: 5-Month Acceptability
Description: as for outcome 3
Time Frame: 5-months
Population: Only intervention participants were asked the items on the System Acceptability Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention
Number analyzed (Participants) | 89
score on a scale | 15.55 (3.15)

5. Secondary Outcome: 3-Month Retention
Description: The retention rate will be calculated based on how many participants in the intervention group have completed the follow-up surveys. A total retention score (those retained/those enrolled) will be computed based on interaction with the WebApp.
Time Frame: 3-months
Population: Retention was calculated based on the total number of participants that completed the Baseline survey.
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 122 | 139
Participants
  Completed 3-Month Survey | 93 | 112
  Did not complete 3-Month Survey | 29 | 27

6. Secondary Outcome: 5-Month Retention
Description: as for outcome 5
Time Frame: 5-months
Population: Retention was calculated based on the total number of participants that completed the Baseline survey.
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 122 | 139
Participants
  Completed 5-Month Survey | 89 | 110
  Did not complete 5-Month Survey | 33 | 29

7. Other Pre Specified Outcome: 3-Month Sexual Violence Victimization
Description: The 10-item Sexual Experiences Survey will be used to measure participants' experiences of sexual violence victimization. The revised Sexual Experiences Survey - Short Form Victimization (Koss et al., 2007) includes 10 items that are used to assess the frequency of seven victimization behaviors and then uses three questions to explore the sex of the perpetrator and if the participant believes they were raped. We will be items 1-7 to assess the number of times an individual has experienced victimization over the last 3 months from 0 to 3+ times. The results will be scored as a percentage of participants who have experienced each individual behavior and the percentage who report that they have experienced a rape.
Time Frame: 3-months
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 93 | 112
Participants
  Victimization - Fondled, Kissed, or Rubbed Against: Experienced | 7 | 13
  Victimization - Fondled, Kissed, or Rubbed Against: Did not experience | 86 | 98
  Victimization - Fondled, Kissed, or Rubbed Against: Not Applicable | 0 | 0
  Victimization - Fondled, Kissed, or Rubbed Against: Missing | 0 | 1
  Victimization - Oral Sex: Experienced | 2 | 7
  Victimization - Oral Sex: Did not experience | 91 | 104
  Victimization - Oral Sex: Not Applicable | 0 | 0
  Victimization - Oral Sex: Missing | 0 | 1
  Victimization - Vaginal Sex: Experienced | 1 | 2
  Victimization - Vaginal Sex: Did not experience | 66 | 67
  Victimization - Vaginal Sex: Not Applicable | 26 | 41
  Victimization - Vaginal Sex: Missing | 0 | 2
  Victimization - Anal Sex: Experienced | 1 | 1
  Victimization - Anal Sex: Did not experience | 92 | 109
  Victimization - Anal Sex: Not Applicable | 0 | 0
  Victimization - Anal Sex: Missing | 0 | 2
  Victimization - Attempted Oral Sex: Experienced | 1 | 5
  Victimization - Attempted Oral Sex: Did not experience | 92 | 105
  Victimization - Attempted Oral Sex: Not Applicable | 0 | 0
  Victimization - Attempted Oral Sex: Missing | 0 | 2
  Victimization - Attempted Vaginal Sex: Experienced | 3 | 3
  Victimization - Attempted Vaginal Sex: Did not experience | 64 | 66
  Victimization - Attempted Vaginal Sex: Not Applicable | 26 | 41
  Victimization - Attempted Vaginal Sex: Missing | 0 | 2
  Victimization - Attempted Anal Sex: Experienced | 1 | 3
  Victimization - Attempted Anal Sex: Did not experience | 92 | 107
  Victimization - Attempted Anal Sex: Not Applicable | 0 | 0
  Victimization - Attempted Anal Sex: Missing | 0 | 2
  Victimization - Rape: Experienced | 2 | 3
  Victimization - Rape: Did not experience | 91 | 107
  Victimization - Rape: Not Applicable | 0 | 0
  Victimization - Rape: Missing | 0 | 2

8. Other Pre Specified Outcome: 5-Month Sexual Violence Victimization
Description: The 10-item Sexual Experiences Survey will be used to measure participants' experiences of sexual violence victimization. The revised Sexual Experiences Survey - Short Form Victimization (Koss et al., 2007) includes 10 items that are used to assess the frequency of seven victimization behaviors and then uses three questions to explore the sex of the perpetrator and if the participant believes they were raped. We will be items 1-7 to assess the number of times an individual has experienced victimization over the last 5 months from 0 to 3+ times. The results will be scored as a percentage of participants who have experienced each individual behavior and the percentage who report that they have experienced a rape.
Time Frame: 5-months
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 89 | 110
Participants
  Victimization - Fondled, Kissed, or Rubbed Against: Experienced | 7 | 10
  Victimization - Fondled, Kissed, or Rubbed Against: Did not experience | 82 | 99
  Victimization - Fondled, Kissed, or Rubbed Against: Not Applicable | 0 | 0
  Victimization - Fondled, Kissed, or Rubbed Against: Missing | 0 | 1
  Victimization - Oral Sex: Experienced | 0 | 0
  Victimization - Oral Sex: Did not experience | 89 | 109
  Victimization - Oral Sex: Not Applicable | 0 | 0
  Victimization - Oral Sex: Missing | 0 | 1
  Victimization - Vaginal Sex: Experienced | 2 | 0
  Victimization - Vaginal Sex: Did not experience | 62 | 68
  Victimization - Vaginal Sex: Not Applicable | 25 | 40
  Victimization - Vaginal Sex: Missing | 0 | 2
  Victimization - Anal Sex: Experienced | 0 | 0
  Victimization - Anal Sex: Did not experience | 89 | 108
  Victimization - Anal Sex: Not Applicable | 0 | 0
  Victimization - Anal Sex: Missing | 0 | 2
  Victimization - Attempted Oral Sex: Experienced | 3 | 5
  Victimization - Attempted Oral Sex: Did not experience | 86 | 103
  Victimization - Attempted Oral Sex: Not Applicable | 0 | 0
  Victimization - Attempted Oral Sex: Missing | 0 | 2
  Victimization - Attempted Vaginal Sex: Experienced | 3 | 3
  Victimization - Attempted Vaginal Sex: Did not experience | 61 | 65
  Victimization - Attempted Vaginal Sex: Not Applicable | 25 | 40
  Victimization - Attempted Vaginal Sex: Missing | 0 | 2
  Victimization - Attempted Anal Sex: Experienced | 0 | 0
  Victimization - Attempted Anal Sex: Did not experience | 89 | 108
  Victimization - Attempted Anal Sex: Not Applicable | 0 | 0
  Victimization - Attempted Anal Sex: Missing | 0 | 2
  Victimization - Rape: Experienced | 3 | 2
  Victimization - Rape: Did not experience | 86 | 106
  Victimization - Rape: Not Applicable | 0 | 0
  Victimization - Rape: Missing | 0 | 2

9. Other Pre Specified Outcome: 3-Month Sexual Violence Perpetration
Description: The 10-item Sexual Experiences Survey will be used to measure participants' experiences of sexual violence perpetration. The revised Sexual Experiences Survey - Short Form Perpetration (Koss et al., 2007) includes seven items that are used to assess the frequency of perpetration of sexual violence behaviors and three questions that explore the sex of the victims and if the individual believes they have perpetrated a rape. We will be using these to assess the number of times an individual has perpetrated sexual violence over the last 3 months from 0 to 3+ times. The results will be scored as a percentage of participants who have perpetrated each individual behavior and the percentage who believe they have perpetrated a rape.
Time Frame: 3-months
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 93 | 112
Participants
  Perpetration - Fondled, Kissed, or Rubbed Against: Perpetrated | 0 | 3
  Perpetration - Fondled, Kissed, or Rubbed Against: Did not perpetrate | 93 | 107
  Perpetration - Fondled, Kissed, or Rubbed Against: Missing | 0 | 2
  Perpetration - Oral Sex: Perpetrated | 0 | 0
  Perpetration - Oral Sex: Did not perpetrate | 93 | 110
  Perpetration - Oral Sex: Missing | 0 | 2
  Perpetration - Vaginal Sex: Perpetrated | 0 | 0
  Perpetration - Vaginal Sex: Did not perpetrate | 93 | 110
  Perpetration - Vaginal Sex: Missing | 0 | 2
  Perpetration - Anal Sex: Perpetrated | 0 | 1
  Perpetration - Anal Sex: Did not perpetrate | 93 | 109
  Perpetration - Anal Sex: Missing | 0 | 2
  Perpetration - Attempted Oral Sex: Perpetrated | 0 | 1
  Perpetration - Attempted Oral Sex: Did not perpetrate | 93 | 109
  Perpetration - Attempted Oral Sex: Missing | 0 | 2
  Perpetration - Attempted Vaginal Sex: Perpetrated | 0 | 0
  Perpetration - Attempted Vaginal Sex: Did not perpetrate | 93 | 110
  Perpetration - Attempted Vaginal Sex: Missing | 0 | 2
  Perpetration - Attempted Anal Sex: Perpetrated | 0 | 0
  Perpetration - Attempted Anal Sex: Did not perpetrate | 93 | 110
  Perpetration - Attempted Anal Sex: Missing | 0 | 2
  Perpetration - Rape: Perpetrated | 0 | 0
  Perpetration - Rape: Did not perpetrate | 93 | 109
  Perpetration - Rape: Missing | 0 | 3

10. Other Pre Specified Outcome: 5-Month Sexual Violence Perpetration
Description: The 10-item Sexual Experiences Survey will be used to measure participants' experiences of sexual violence perpetration. The revised Sexual Experiences Survey - Short Form Perpetration (Koss et al., 2007) includes seven items that are used to assess the frequency of perpetration of sexual violence behaviors and three questions that explore the sex of the victims and if the individual believes they have perpetrated a rape. We will be using these to assess the number of times an individual has perpetrated sexual violence over the last 5 months from 0 to 3+ times. The results will be scored as a percentage of participants who have perpetrated each individual behavior and the percentage who believe they have perpetrated a rape.
Time Frame: 5-months
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 89 | 110
Participants
  Perpetration - Fondled, Kissed, or Rubbed Against: Perpetrated | 1 | 1
  Perpetration - Fondled, Kissed, or Rubbed Against: Did not perpetrate | 88 | 108
  Perpetration - Fondled, Kissed, or Rubbed Against: Missing | 0 | 1
  Perpetration - Oral Sex: Perpetrated | 0 | 1
  Perpetration - Oral Sex: Did not perpetrate | 89 | 108
  Perpetration - Oral Sex: Missing | 0 | 1
  Perpetration - Vaginal Sex: Perpetrated | 0 | 0
  Perpetration - Vaginal Sex: Did not perpetrate | 89 | 109
  Perpetration - Vaginal Sex: Missing | 0 | 1
  Perpetration - Anal Sex: Perpetrated | 0 | 0
  Perpetration - Anal Sex: Did not perpetrate | 89 | 109
  Perpetration - Anal Sex: Missing | 0 | 1
  Perpetration - Attempted Oral Sex: Perpetrated | 0 | 0
  Perpetration - Attempted Oral Sex: Did not perpetrate | 89 | 109
  Perpetration - Attempted Oral Sex: Missing | 0 | 1
  Perpetration - Attempted Vaginal Sex: Perpetrated | 2 | 0
  Perpetration - Attempted Vaginal Sex: Did not perpetrate | 87 | 109
  Perpetration - Attempted Vaginal Sex: Missing | 0 | 1
  Perpetration - Attempted Anal Sex: Perpetrated | 0 | 0
  Perpetration - Attempted Anal Sex: Did not perpetrate | 89 | 109
  Perpetration - Attempted Anal Sex: Missing | 0 | 1
  Perpetration - Rape: Perpetrated | 0 | 0
  Perpetration - Rape: Did not perpetrate | 89 | 109
  Perpetration - Rape: Missing | 0 | 1

11. Other Pre Specified Outcome: 3-Month Sexual Violence Knowledge
Description: An 8-item (investigator created) scale will be used to measure participants' sexual violence knowledge at 3-months. The investigator-created sexual violence knowledge questions are scored from 1 (Strongly Agree) to 5 (Strongly Disagree) and the scores will be reverse-coded and summed for a total sexual violence knowledge score ranging from 8 - 40, with higher scores indicating more sexual violence knowledge.
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 93 | 112
score on a scale | 35.81 (3.67) | 36.61 (4.64)

12. Other Pre Specified Outcome: 5-Month Sexual Violence Knowledge
Description: An 8-item (investigator created) scale will be used to measure participants' sexual violence knowledge at 5-months. The investigator-created sexual violence knowledge questions are scored from 1 (Strongly Agree) to 5 (Strongly Disagree) and the scores will be reverse-coded and summed for a total sexual violence knowledge score ranging from 8 - 40, with higher scores indicating more sexual violence knowledge.
Time Frame: 5-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 89 | 110
score on a scale | 35.72 (3.54) | 36.67 (5.10)

13. Other Pre Specified Outcome: 3-Month Sexual Relationship Power
Description: Fifteen items from the Relationship Control sub-scale of the Sexual Relationship Power Scale will be used to measure power dynamics within participants' sexual relationships at 3-months. The Relationship Control Sub-scale Items (Pulerwitz, Gortmaker, & DeJong, 2000) are scored from 1 (Strongly Agree) to 4 (Strongly Disagree). Scores are summed with total scores ranging from 15-60. Higher scores represent higher sexual relationship power.
Time Frame: 3-months
Population: Only participants who chose a relationship status other than "Single" were asked the SRPS questions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 29 | 34
score on a scale | 49.34 (6.03) | 50.53 (6.16)

14. Other Pre Specified Outcome: 5-Month Sexual Relationship Power
Description: Fifteen items from the Relationship Control sub-scale of the Sexual Relationship Power Scale will be used to measure power dynamics within participants' sexual relationships at 5-months. The Relationship Control Sub-scale Items (Pulerwitz, Gortmaker, & DeJong, 2000) are scored from 1 (Strongly Agree) to 4 (Strongly Disagree). Scores are summed with total scores ranging from 15-60. Higher scores represent higher sexual relationship power.
Time Frame: 5-months
Population: Only participants who chose a relationship status other than "Single" were asked the SRPS questions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 27 | 42
score on a scale | 50.56 (6.20) | 51.55 (5.62)

15. Other Pre Specified Outcome: 3-Month Rape Myth Acceptance
Description: The 22-item modified Illinois Rape Myth Acceptance scale will be used to measure attitudes endorsing rape myths at 3-months. The modified Illinois Rape Myth Acceptance Scale (McMahon & Farmer, 2011) is scored from 1 (Strongly Agree) to 5 (Strongly Disagree). It includes four sub-scales (She asked for it, He didn't mean to, It wasn't really rape, and She lied). The items in each sub-scale can be summed for a total score and the scores for the entire scale can be summed for a cumulative score. Scores on the full scale range from 22-110. Scores on the She Asked For It and He Didn't Mean To sub-scales range from 6-30. Scores on the It Wasn't Really Rape and the She Lied sub-scales range from 5-25. Higher scores indicate greater rejection of rape myths.
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 93 | 112
score on a scale
  Full Scale | 95.33 (12.57) | 93.98 (15.48)
  She Asked for It Sub-scale | 26.17 (3.98) | 26.49 (4.51)
  He Didn't Mean To Sub-scale | 24.06 (4.27) | 23.66 (5.02)
  It Wasn't Really Rape Sub-scale | 23.45 (2.76) | 22.88 (3.73)
  She Lied Sub-scale | 21.65 (3.72) | 20.95 (4.56)

16. Other Pre Specified Outcome: 5-Month Rape Myth Acceptance
Description: The 22-item modified Illinois Rape Myth Acceptance scale will be used to measure attitudes endorsing rape myths at 5-months. The modified Illinois Rape Myth Acceptance Scale (McMahon & Farmer, 2011) is scored from 1 (Strongly Agree) to 5 (Strongly Disagree). It includes four sub-scales (She asked for it, He didn't mean to, It wasn't really rape, and She lied). The items in each sub-scale can be summed for a total score and the scores for the entire scale can be summed for a cumulative score. Scores on the full scale range from 22-110. Scores on the She Asked For It and He Didn't Mean To sub-scales range from 6-30. Scores on the It Wasn't Really Rape and the She Lied sub-scales range from 5-25. Higher scores indicate greater rejection of rape myths.
Time Frame: 5-months
Population: One participant from the Control group had missing data and was not included in data analysis for the Rape Myth Acceptance measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 89 | 109
score on a scale
  Full Scale | 96.08 (10.20) | 96.30 (12.86)
  She Asked for It Sub-scale | 26.60 (3.80) | 26.80 (3.94)
  He Didn't Mean To Sub-scale | 24.00 (3.98) | 24.69 (4.50)
  It Wasn't Really Rape Sub-scale | 23.58 (2.09) | 23.29 (2.70)
  She Lied Sub-scale | 21.90 (3.35) | 21.52 (3.77)

ADVERSE EVENTS:
Time Frame: 5 months
Description: Since this was an anonymous study, adverse events were defined as those reported to study staff.
Arm/Group | MKit WebApp Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/139
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/139
Other Adverse Events (participants affected / at risk) | 0/122 | 0/139

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT03316911/Prot_SAP_000.pdf